CLINICAL TRIAL: NCT04720872
Title: Manual Therapy Combined With Physical Therapist-Directed Vestibular Rehabilitation in Patients With Unilateral Peripheral Vestibular Hypofunction: A Randomized Controlled Trial.
Brief Title: Manual Therapy With Directed Vestibular Rehabilitation in Patients With Unilateral Peripheral Vestibular Hypofunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén.
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Vestibular Disorder
Keywords: Manual therapy; vestibular rehabilitation; unilateral peripheral vestibular hypofunction; Dizziness; balance confidence; postural control.
MeSH Terms: conditions — Dizziness | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): * Manual therapy: 4 sessions, 1 session per week (20 minutes approximately).
  * Physical therapist-directed vestibular rehabilitation: 4 weeks, 1 session per week with the physical therapist (30 minutes approximately), after manual therapy.
  * Home based vestibular rehabilitation: 4 weeks (2 sessions per day).
  Interventions: Other: Manual therapy and vestibular rehabilitation treatment
- Control group (No Intervention): Home based vestibular rehabilitation: 4 weeks (2 sessions per day). The participants attended the center once a week to check correct execution of the exercises.

INTERVENTIONS:
Other: Manual therapy and vestibular rehabilitation treatment — The experimental group received manual therapy and vestibular rehabilitation treatment.
  Arms: Experimental group

SUMMARY:
Randomized clinical trial with a control group that aims to evaluate the effects of a manual therapy protocol, together with a physical therapist-directed vestibular rehabilitation program, in patients with unilateral peripheral vestibular hypofunction. The intervention period will last approximately 4 weeks. Outcome measures will be collected at baseline, just after the intervention, as well as 1 and 6 months after the intervention.

DETAILED DESCRIPTION:
Peripheral vestibular disorders are common in otorhinolaryngology practice. These patients often complain of vertigo and dizziness, as well as balance problems, causing an important impact on health-related quality of life. The objective of this study was to investigate the effects of manual therapy combined with physical therapist-directed vestibular rehabilitation in patients with unilateral peripheral vestibular hypofunction. The design of this study is a randomized controlled trial with two groups (experimental and control groups). The impact of dizziness on daily function and quality of life (Dizziness Handicap Inventory), the fear of falling and the balance confidence (Activities-specific Balance Confidence scale-16 items), postural control (stabilometric platform) as well as the intensity (visual analogue scale) and number of the vertiginous crisis will be determined. The intervention period will last four weeks. Participants of the experimental group will receive 4 sessions of manual therapy together with physical therapist-directed vestibular rehabilitation, while participants of the control group will receive home-based vestibular rehabilitation. Outcome measurements will take place at baseline, immediately after the intervention, one month and six months after the intervention. Within-group and between-group data will be analyzed and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with a clinical diagnosis of unilateral peripheral vestibular hypofunction confirmed by Video Head Impulse Test (< 0.8), referring balance impairments, postural instability, gait instability, vertigo, dizziness or motion sensitivity, able to understand and complete e instructions, programs, and protocols of this project, and providing a signed informed consent.

Exclusion Criteria:

* Central nervous system, degenerative or cancer diseases, acute infection.
* Morphological/ functional alterations of the lower limbs, and/or morphological alteration of the cervical and/or suboccipital rachis.
* Conditions (i.e. neuromuscular disease or traumatism) that contraindicate the performance of the exercises and interventions of this study, as well as cognitive impairment that prevents the participants from understanding and completing the questionnaires and interventions.
* Positive results for the Klein test and the Rancurel test, or cerebrovascular alterations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | Baseline-4 weeks
  Evaluates the level of disability related to the impact of dizziness on daily function and quality of life.

SECONDARY OUTCOMES:
ABC-16 (Activities-specific Balance Confidence scale-16 ítems) | Baseline-4 weeks
  Questionnaire that assesses balance confidence in performing activities of daily living.
STABILOMETRIC PLATFORM | Baseline-4 weeks
  Instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
Visual-Analogue-Scale (VAS) | Baseline-4 weeks
  The intensity of the vertiginous crisis will be assessed by a visual-analogue-scale during the 4 weeks of the intervention period, respectively.
The number of crisis | Baseline-4 weeks
  The frequency of the vertiginous crisis will be assessed by the number of crisis during the 4 weeks of the intervention period, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Ciudad de Jaén. Av. del Ejército Español, 10, 23007; University of Jaén. Campus Las Lagunillas s/n. 23071, Jaén, Spain